CLINICAL TRIAL: NCT03399890
Title: The Influence of Neuromuscular Reversal With Neostigmine or Sugammadex on Neurological Physical Exam Time in Lumbar Neurosurgical Cases.
Brief Title: The Influence of Neuromuscular Reversal on Neurological Physical Exam Time in Lumbar Neurosurgical Cases.
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Basak Ceyda MECO, Associate Prof., Ankara University
Other Study IDs: 10-544
Record Dates: First submitted 2017-12-11; First posted 2018-01-17 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Neurological Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group S: Group S: Group sugammadex Patients in this group received sugammadex at the end of the surgery, as neuromuscular reversal agent. Neurological physical exam time was recorded.
  Interventions: Diagnostic Test: Neurological physical exam
- Group N: Group N: Group Neostigmine
  Patients in this group received neostigmine at the end of the surgeryas neuromuscular reversal agent. Neurological physical exam time was recorded.
  Interventions: Diagnostic Test: Neurological physical exam

INTERVENTIONS:
Diagnostic Test: Neurological physical exam — Neurological physical exam is performed in all patients at the OR table, immediately after the operation.

SUMMARY:
Neurological physical exam is a very important outcome that should be evaluated as soon as possible after every lumbar procedures. The aim of this study was to evaluate the neurological physical examination time after lumbar procedures.

DETAILED DESCRIPTION:
Neurological physical exam is a very important outcome that should be evaluated as soon as possible after every lumbar procedures. By that early postoperative neurological complications can be revealed and early interventions planned. The aim of this study was to evaluate the neurological physical examination time after lumbar procedures. Two routinely used different reversal agents (neostigmine or sugammadex) were compared according reversal times and muscle strength on PACU admission.

ELIGIBILITY:
Inclusion Criteria:

* Lumber surgery
* ASA I-II
* Elective surgery

Exclusion Criteria:

* Emergency cases
* Age lower than 18
* Age higher than 65
* Patient with existing neurological deficit
* Patient with existing renal insufficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All lumbar surgeries performed during the study period were enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Neurological physical examination time | postoperative first 30 minutes
  Neurological physical examination time

SECONDARY OUTCOMES:
Muscle strength at PACU transfer | postoperative first 60 minutes
  Muscle strength at PACU transfer (evaluated with a 5 point scale) 0/5: no contraction in muscles 1/5: muscle flicker but no movement 2/5: movement possible bıt not against gravity (test the joint in its horizontal plane) 3/5: moment possible against gravity but not against resistance by the examiner 4/5: movement possible against resistance by the examiner 5/5: normal strength

CONTACTS AND LOCATIONS:
Overall Officials: Basak Ceyda MECO, MD, Principal Investigator — Ankara University Faculty of Medicine
Locations (1):
- Ankara University Faculty of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No